CLINICAL TRIAL: NCT05604729
Title: The Effect on Envelope of Motion in Asymptomatic Bruxers - A Double Blinded Study
Brief Title: The Effect on Envelope of Motion in Asymptomatic Bruxers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Region Västerbotten (Other Government)
Collaborators: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BoNT A - Morphology
Record Dates: First submitted 2022-04-01; First posted 2022-11-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Tooth Wear; Bruxism
MeSH Terms: conditions — Tooth Wear; Bruxism | interventions — Botulinum Toxins, Type A; incobotulinumtoxinA; Isotonic Solutions

STUDY DESIGN:
Intervention Model Description: Double blinded
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Computerised randomisation, colour coded intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- BoNT A (botulinum neurotoxin type A) (Experimental): Botulinum neurotoxin, 25 units (U) into each masseter at three sessions.
  Interventions: Drug: Botulinum toxin type A
- Placebo (Placebo Comparator): Saline solution
  Interventions: Drug: Placebo
- Control (Placebo Comparator): Saline solution, no tooth wear
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Botulinum toxin type A — Botulinum Neurotoxin type A
  Other Names: Xeomin
  Arms: BoNT A (botulinum neurotoxin type A)
Drug: Placebo — Saline solution
  Other Names: Isotonic solution
  Arms: Control; Placebo

SUMMARY:
Investigating the effect of botulinum neurotoxin on the jaw-neck envelope of motion.

DETAILED DESCRIPTION:
Research subjects will be allocated to placebo or botulinum neurotoxin intervention. A control group will not receive any intervention. The intervention will be administered at three separate sessions with 12 weeks in between. Prior to intervention, and 6 months after last intervention the jaw-neck envelope of motion will be studied using 3D optoelectronic recording systems.

ELIGIBILITY:
Inclusion Criteria:

• Tooth wear into dentin.

Exclusion Criteria:

* No temporomandibular pathology.
* No drugs affecting the central nervous system.
* No conditions affecting muscles or central nervous system.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of range of motion | Baseline and 6 months after last intervention. Measurements compared to baseline values.
  Measured on a cartesian plane in millimeters.
Change of envelope of motion | Baseline and 6 months after last intervention. Measurements compared to baseline values.
  Volume of envelope of motion measured in cubic millimeters.
Change of length in chewing cycles | Baseline and 6 months after last intervention. Measurements compared to baseline values.
  Repetitive chewing cycles, measured in milliseconds.

SECONDARY OUTCOMES:
Change of muscle thickness | Baseline and 6 months, 1 year and 2 years after last intervention. Measurements compared to baseline values.
  Masseter muscle thickness measured through ultrasonography
Change of maximal voluntary bite force | Baseline and 6 months, 1 year and 2 years after last intervention. Measurements compared to baseline values.
  Measured through a strain gauge meter
Tooth wear, change of hard tissue mass | Baseline and 6 months, 1 year and 2 years after last intervention. Measurements compared to baseline values.
  Intraoral scanning. Tooth wear measured in cubic millimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Pettersson, PhD, Principal Investigator — Umeå University
Locations (1):
- Norrlands universitetssjukhus, Umeå, Västerbotten County, Sweden

IPD SHARING:
Plan to Share IPD: No